CLINICAL TRIAL: NCT06598995
Title: The Association Between Myocardial Bridging and Atrial Fibrillation in Patients With Obstructive Hypertrophic Cardiomyopathy
Brief Title: Myocardial Bridging in Obstructive Hypertrophic Cardiomyopathy
Acronym: MB in oHCM
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Changrong Nie, MD, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2022-1892; 2022-GSP-GG-29 (Other Grant/Funding Number: National High Level Hospital Clinical Research Funding)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myocardial Bridging; Obstructive Hypertrophic Cardiomyopathy; Atrial Fibrillation (AF)
MeSH Terms: conditions — Myocardial Bridging; Cardiomyopathy, Hypertrophic; Atrial Fibrillation | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstructive hypertrophic cardiomyopathy who underwent septal myectomy: All patients underwent angiography and without other coronary artery disease.
  Interventions: Procedure: Coronary artery bypass grafting or unroofing

INTERVENTIONS:
Procedure: Coronary artery bypass grafting or unroofing — Patients had an MB with >75% compression degree would receive coronary artery bypass grafting, and those who underwent unroofing may had a depth of MB < 5mm (whether deal with these MB with a depth <5mm depends on the surgeon and the period time of patients received a surgery).

SUMMARY:
This study investigated the impact of myocardial bridging (MB) and its characteristics on preoperative atrial fibrillation and survival in patients with obstructive hypertrophic cardiomyopathy (oHCM). We recruited 968 consecutive patients with oHCM who underwent myectomy at our institution between January 2015 and December 2019, including 144 patients with MB and 824 patients without MB. All patients received angiography before surgery. The diagnosis of preoperative atrial fibrillation was based on 12-lead electrocardiography, 24-hour Holter electrocardiography, or in-hospital electrocardiogram monitoring, which was extracted from patients' medical records. Surgical details and follow-up data were also collected.

ELIGIBILITY:
Inclusion Criteria:I(i) age ≥ 18 years and (ii) diagnosis of oHCM based on clinical and echocardiographic evaluation.

-

Exclusion Criteria: (i) a history of heart surgery (ii) Patients who had coronary atherosclerosis or myocardial infraction; (iii) Patients who had no angiography records.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients diagnosed with obstructive hypertrophic cardiomyopathy who underwent septal myectomy.
Sampling Method: Probability Sample
Enrollment: 968 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause death | One month after discharge
  Any death occurred one month after discharge

SECONDARY OUTCOMES:
New-onset AF | One month after discharge.
  Patients did not have AF before surgery, and AF occurred one month after discharge.
Composite endpoints | One month after discharge
  Composite endpoints including all-cause death, new-onset AF, and readmission due to heart failure, stroke, and other cardiovascular events (such as myocardial infarction, arrhythmia).

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Please Select, China

IPD SHARING:
Plan to Share IPD: No